CLINICAL TRIAL: NCT05300932
Title: Efficacy and Safety of Baricitinib in Systemic Sclerosis: a Phase IV, Double-blinded, Controlled Study.
Brief Title: A Study Evaluating the Efficacy and Safety of Baricitinib in Systemic Sclerosis
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Eli Lilly and Company (Industry); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, YIKAI YU, Clinical Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-SSc202203
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis，Baricitinib
MeSH Terms: conditions — Scleroderma, Systemic | interventions — baricitinib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baricitinib 4mg (Experimental): 4mg of oral Baricitinib everyday for 48 weeks.
  Interventions: Drug: Baricitinib
- Cyclophosphamide (Active Comparator): Subject received cyclophosphamide 400mg intravenous drip every 2 weeks combined with oral Prednisone 10-15 mg/d （standard of care）through the 24 weeks double blind period. Subsequently, subject were administered oral Baricitinib 4mg everyday through the 24-48 weeks open label period.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Baricitinib — Orally take Baricitinib 4mg everyday for 48 weeks
  Other Names: Olumiant
  Arms: Baricitinib 4mg
Drug: Cyclophosphamide — Subject received cyclophosphamide 400mg intravenous drip every 2 weeks combined with oral Prednisone 10-15 mg/d （standard of care）through the 24 weeks double blind period. Subsequently, subject were administered oral Baricitinib 4mg everyday through the 24-48 weeks open label period.
  Other Names: Cytoxan
  Arms: Cyclophosphamide

SUMMARY:
Systemic Sclerosis (Ssc) is a rare, systemic autoimmune disease characterized by skin fibrosis and vasculopathy. In addition to the skin, it is a heterogeneous disease that affects multiple organs, including the musculoskeletal, cardiac, pulmonary, and gastrointestinal systems. Patients may experience many symptoms such as pain, fatigue, dyspnea, impaired hand function, dry mouth, and difficulty sleeping. As a result of these symptoms, these patients may experience a decrease in activities of daily living, physical activity level and quality of life, while psychological problems such as anxiety and depression may increase.

DETAILED DESCRIPTION:
This is a 48 weeks, prospective, double-blind, controlled study. The specific objectives of this study are to:

1. Determine whether Baricitinib is effective and safe in the treatment of patients with diffuse cutaneous (dc)SSc when compared to patients treated with CTX. In this study, stand of care of GC is permitted to use.
2. Determine whether Baricitinib is more effective than CTX, as measured by change in CRISS, which is a composite outcome measure provisionally endorsed by the ACR for scleroderma clinical trials. It incorporates change in the mRSS, FVC percent predicted, physician and patient global assessments, and HAQ-DI. Additionally, hemoglobin corrected diffusion capacity (DLCO), Medsger Severity Scale (MSS), and by other physician and patient derived outcome measures will be used.
3. Determine the biological activity of Baricitinib vs CTX as assessed by effect on histology of skin, gene expression of skin and blood, change in B-Cell profiles including assessment of B regulatory cells, and effect on serological and cutaneous biomarkers of disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Systematic Sclerosis (SSc), as defined using the 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc
2. Diffuse Systemic Sclerosis (dcSSc) as defined by LeRoy and Medsger
3. Disease duration of ≤ 36 months (defined as time from the first non-Raynaud phenomenon manifestation)
4. For disease duration of ≤ 18 months: ≥ 10 and ≤ 35 mRSS units at the screening visit
5. For disease duration of >18-36 months: ≥ 15 and ≤ 45 mRSS units at the screening visit and one of the following:

1)Increase ≥ 3 in mRSS units compared with the last visit within previous 1-6 months 2)Involvement of one new body area with ≥ 2 mRSS units compared with the last visit within the previous 1-6 months 3)Involvement of two new body areas with ≥ 1 mRSS units compared with the last visit within the previous 1-6 months 4)Presence of 1 or more Tendon Friction Rub 6.Age ≥ 18 years at the screening visit 7.If female of childbearing potential, the patient must have a negative pregnancy test at screening and baseline visits 8.Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) and NSAIDs are permitted if the patient is on a stable dose regimen for 2 weeks prior to and including the baseline visit.

9.ACE inhibitors, calcium-channel blockers, proton-pump inhibitors, and/or oral vasodilators are permitted if the patient is on a stable dose for ≥ 2 weeks prior to and including the baseline visit.

Exclusion Criteria:

1. Rheumatic disease other than dcSSc; it is acceptable to include patients with fibromyalgia and scleroderma-associated myopathy
2. Limited cutaneous systemic sclerosis or sine scleroderma at the screening visit
3. Major surgery (including joint surgery) within 8 weeks prior to screening visit
4. Infected ulcer prior to treatment
5. Treatment with any investigational agent within ≤ 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of the baseline visit
6. Previous treatment with cell-depleting therapies, including investigational agents, including but not limited to, CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19, and ABA
7. Anti-CD20 within 12 months prior to baseline visit.
8. Use of Intravenous Immunoglobulin (IVIG) within 12 weeks prior to baseline visit
9. Previous treatment with chlorambucil, bone marrow transplantation, or total lymphoid irradiation
10. Immunization with a live/attenuated vaccine within ≤ 4 weeks prior to the baseline visit
11. Treatment with methotrexate, hydroxychloroquine, cyclosporine A, azathioprine, mycophenolate mofetil rapamycin, colchicine, or D-penicillamine, within≤ 4 weeks prior to the baseline visit
12. Treatment with etanercept within ≤ 2 weeks, infliximab, certolizumab, golimumab, ABA or adalimumab within ≤ 8 weeks, anakinra within ≤ 1 week prior to the baseline visit
13. Pulmonary disease with FVC ≤ 50% of predicted, or DLCO (uncorrected for hemoglobin ) ≤ 40% of predicted at the screening visit
14. Pulmonary arterial hypertension (PAH) as determined by right heart catheterization or on PAH approved medications for PAH. It is acceptable to use PDFE-5 inhibitors for Raynaud's and digital ulcers.
15. Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be participants with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
16. Positive for hepatitis B surface antigen prior to the baseline visit
17. Positive for hepatitis C antigen, if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay prior to baseline visit
18. Subjects at risk for tuberculosis (TB). Specifically excluded from this study will be participants with a history of active TB within the last 3 years, even if it was treated; a history of active TB greater than 3 years ago, unless there is documentation that the prior anti-TB treatment was appropriate in duration and type; current clinical, radiographic, or laboratory evidence of active TB; and latent TB that was not successfully treated (≥ 4 weeks).
19. Any of the following at the screening visit: Hemoglobin <8 g/dL; ANC < 1,000/mm3 (<1 x 109/L); platelets < 100,000/mm3 (<100 x 109/L); serum creatinine > 2 x ULN; serum ALT or AST > 2 x ULN
20. Severe skin thickening (mRSS 3) on the inner aspects of thighs, upper arms, or abdomen
21. Patients with a history of anaphylaxis to Baricitinib or cyclophosphamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified Rodnan skin score (mRSS) at week 24 | 24 weeks
  Change in modified Rodnan skin score (mRSS) at week 24 performed by the same investigator at week 0 and week 24 and the change in mRSS will be calculated following the formula: ΔmRSS= mRSSw24 - mRSSw0.
  To measure mRSS, skin thickness of the patient is rated by palpation at each of 17 anatomic sites using a scale of 0-3 (0 = normal skin; 1= mild thickness; 2= moderate thickness; 3=severe thickness with an inability to pinch the skin into a fold). The scores at each site are summed with a minimum of 0 and a maximum of 51 (17 sites)

SECONDARY OUTCOMES:
Incidence of death | 24 & 48 weeks
  Incidence of death
Incidence of Adverse Events | 24 & 48 weeks
  according to the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading scale
Incidence of Severe Adverse Events | 24 & 48 weeks
  according to the Common Terminology Criteria for Adverse Events (CTCAE) toxicity grading scale
Change in modified Rodnan skin score at 12，24，32，40，48 weeks | 12，24，32，40，48 weeks
  Change in modified Rodnan skin score at 12，24，32，40，48 weeks
Proportion of patients who improved mRSS at 12，24，32，40，48 weeks | 12，24，32，40，48 weeks
  Proportion of patients who improved mRSS at 12，24，32，40，48 weeks
Proportion of patients with an active disease according to the European scleroderma trials and research group (EUSTAR)SSc activity score at 12，24，48 weeks | 12，24，32，40，48 weeks
  EUSTAR SSc activity index score from 0 to 10 - a cut-off ≥ 2.5 identifies patients with active disease
Change in the Combined Response Index in Diffuse Systemic Sclerosis (CRISS) score | 24，48 weeks
  composite response index
SSc disease activity | 12，24，32，40，48 weeks
  Physicians visual analogue scale range from 0 (min) to 10 (max) - 0=no activity, 10=maximum activity Patients visual analogue scale range from 0 (min) to 10 (max) - 0=no activity, 10=maximum activity
Short Form-36 (SF-36) health questionnaire | 0, 12，24，32，40，48 weeks
  self-administered questionnaire of 36 items assessing the following 8 domains : physical functioning, bodily pain, role limitations attributable to physical health problems, general health perceptions, mental health, role limitations to emotional problems, vitality and social functioning (scale from 0 to 100)
EurolQol-5Domain (EQ-5D) health questionnaire | 0, 12，24，32，40，48 weeks
  self reported measure of quality of life - (scale from 0 to 100)
Health Assessment Questionnaire Disability Index (HAQ-DI) scale | 0, 12，24，32，40，48 weeks
  self administered 20 questions- score range from 0 (no disability) to 3 (severe disability)

CONTACTS AND LOCATIONS:
Overall Officials: AIHUA DU, Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - Department of RheumatologyTongji Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No